CLINICAL TRIAL: NCT02295514
Title: Correlation Between PTP1B Expression and Organ Failure During Sepsis
Acronym: SEPP1B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2014/087/HP
Record Dates: First submitted 2014-10-23; First posted 2014-11-20 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Sepsis
Keywords: Sepsis; Septic shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PTP1B dosage (Experimental): PTP1B dosage during sepsis
  Interventions: Biological: PTP1B dosage

INTERVENTIONS:
Biological: PTP1B dosage — PTP1B sampled and dosed during sepsis

SUMMARY:
Despite major advances in the treatment and understanding of the pathophysiological mechanisms, mortality of severe sepsis remains high, ranging from 25 to 50%. With a prevalence > 20% in intensive care units, it is now in a population increasingly aging with many co-morbidities, a real public health problem. Thus, changes in treatment to physiological axes could change the prognosis of these patients. Protein Tyrosine Phosphatase 1B (PTP1B) is involved in the negative regulation of many cellular pathways such as the response to insulin, leptin and certain growth factors and endothelial nitric oxide production. PTP1B appears to be particularly involved in the control of endothelial function and insulin secretion. Under these conditions, encouraging results have been obtained in a model of insulin resistance (obesity, diabetes) and as part of pro-angiogenic therapy by inhibition of PTP1B on models of heart failure. Recent advances have broadened the pathophysiological implications of PTP1B conferring a potential role in the regulation of inflammatory processes. In an experimental model of septic shock (Inserm 1096), the investigators demonstrated a significant improvement in survival and cardiovascular function in genetically deficient mice PTP1B (PTP1B - / -). Finally, PTP1B is involved in the downregulation of the signaling pathway of insulin via a feedback phenomenon. Septic shock induces many changes in carbohydrate metabolism. These changes result in hyperglycemia associated with insulin resistance, an independent risk factor of morbidity and mortality. Taken together, these data suggest that the expression of PTP1B could be useful in septic patients by modulating insulin resistance and thus the prognosis of these patients. This justifies the investigator clinical research project on the relationship between the expression of PTP1B levels, glycemic status and prognosis evaluated by the SOFA score in patients with septic shock with multiple organ failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients in ICU for septic shock
* Person belonging to a social security system
* Informed patient who signed consent
* Contraceptive method in women of reproductive age

Exclusion Criteria:

* Pregnancy
* Patient not able to take a decision because of an administrative or legal decision
* Patient participating to an other interventional study
* BMI > 30 kg/m2
* Diabetes with specific treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in PTP1B level expression | Day 5
  Change from baseline in PTP1B level expression by biological analysis
Number of patients with organ failure | Day 5
  Number of patients with organ failure

SECONDARY OUTCOMES:
Dose of insulin administered during the sepsis | Day 5
  cumulative dose of insulin administered in the first 5 days of hospitalization
Insulin resistance evaluation | Day 1
  Evaluation of insulin resistance by biological analysis
Blood glucose Analysis | Day 5
  Analysis of the variability in Blood glucose
Number of death participants at ICU discharge | ICU discharge, day 28
  ICU mortality at day 28
Number of death participants at at the end of the study | Day 28
  Mortality at day 28
Number of death participants at at hospital discharge | 10 days (average)
  Mortality at hospital discharge, average of 10 days after surgical intervention
Duration of mechanical ventilation | Day 28
  Duration of mechanical ventilation from admission to discharge

CONTACTS AND LOCATIONS:
Overall Officials: steven grangé, MD, Principal Investigator — Rouen Universitary Hospital
Locations (1):
- Rouen University Hospital, Rouen, France

REFERENCES:
- [Background] Elchebly M, Payette P, Michaliszyn E, Cromlish W, Collins S, Loy AL, Normandin D, Cheng A, Himms-Hagen J, Chan CC, Ramachandran C, Gresser MJ, Tremblay ML, Kennedy BP. Increased insulin sensitivity and obesity resistance in mice lacking the protein tyrosine phosphatase-1B gene. Science. 1999 Mar 5;283(5407):1544-8. doi: 10.1126/science.283.5407.1544. PMID 10066179
- [Background] Coquerel D, Neviere R, Delile E, Mulder P, Marechal X, Montaigne D, Renet S, Remy-Jouet I, Gomez E, Henry JP, do Rego JC, Richard V, Tamion F. Gene deletion of protein tyrosine phosphatase 1B protects against sepsis-induced cardiovascular dysfunction and mortality. Arterioscler Thromb Vasc Biol. 2014 May;34(5):1032-44. doi: 10.1161/ATVBAHA.114.303450. Epub 2014 Feb 27. PMID 24578383
- [Background] Traves PG, Pardo V, Pimentel-Santillana M, Gonzalez-Rodriguez A, Mojena M, Rico D, Montenegro Y, Cales C, Martin-Sanz P, Valverde AM, Bosca L. Pivotal role of protein tyrosine phosphatase 1B (PTP1B) in the macrophage response to pro-inflammatory and anti-inflammatory challenge. Cell Death Dis. 2014 Mar 13;5(3):e1125. doi: 10.1038/cddis.2014.90. PMID 24625984
- [Background] Zabolotny JM, Kim YB, Welsh LA, Kershaw EE, Neel BG, Kahn BB. Protein-tyrosine phosphatase 1B expression is induced by inflammation in vivo. J Biol Chem. 2008 May 23;283(21):14230-41. doi: 10.1074/jbc.M800061200. Epub 2008 Feb 14. PMID 18281274
- [Background] Ali MI, Ketsawatsomkron P, Belin de Chantemele EJ, Mintz JD, Muta K, Salet C, Black SM, Tremblay ML, Fulton DJ, Marrero MB, Stepp DW. Deletion of protein tyrosine phosphatase 1b improves peripheral insulin resistance and vascular function in obese, leptin-resistant mice via reduced oxidant tone. Circ Res. 2009 Nov 6;105(10):1013-22. doi: 10.1161/CIRCRESAHA.109.206318. Epub 2009 Sep 24. PMID 19797171
- [Result] Feldhammer M, Uetani N, Miranda-Saavedra D, Tremblay ML. PTP1B: a simple enzyme for a complex world. Crit Rev Biochem Mol Biol. 2013 Sep-Oct;48(5):430-45. doi: 10.3109/10409238.2013.819830. Epub 2013 Jul 23. PMID 23879520